CLINICAL TRIAL: NCT00000291
Title: Effects of Labetalol on Human Cocaine Use
Brief Title: Effects of Labetalol on Human Cocaine Use - 8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-8; P50-09259-8
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Labetalol

INTERVENTIONS:
Drug: Labetalol

SUMMARY:
The purpose of this study is to determine the effect of labetalol treatment on the subjective and physiological effects of cocaine.

DETAILED DESCRIPTION:
The goal of this study was to investigate the safety and utility of labetalol an alpha and beta adrenergic block, for cocaine dependence in humans. A total of 12 subjects were enrolled in this double blind, placebo controlled outpatient study. After baseline measures are obtained, three experimental sessions were held at least 2 days apart. Subjects were administered a single low (100 mg) or high dose of labetalol (200mg) or placebo on each of 3 experimental sessions. The labetalol doses were given in ascending order and the placebo treatment were randomly inserted into the sequence. A single dose of smoked cocaine (0.4 mg/kg) was administered 2 hrs after labetalol or placebo treatment. During the sessions, several subjective, behavioral and physiological measures were obtained.

ELIGIBILITY:
Inclusion Criteria:

Male/Female ages 20-55. History of smoked or intravenous cocaine use on the average of at least once a week over a six month period. Current history of good health and normal EKG. Not pregnant as determined by pregnancy screening nor breat feeding and using acceptable birth control methods (e.g. birth control pills diaphragm, condoms, plus foam) during the study.

Exclusion Criteria:

Current problems with major psychiatric illnesses including bipolar disorder, schizophrenia, or anxiety disorders. Current dependence on alcohol or on durgs other than cocaine. History of major medical illnesses including asthma and chronic obstructive pulmonary disease. Currently on a drug related parole or probation. Treated for chemical dependency within the past 6 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1997-10; Study Completion 2001-12

PRIMARY OUTCOMES:
Subjective
Physiological measures

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Pharmacol. Biochem. Behav (accepted). None